CLINICAL TRIAL: NCT02015728
Title: The Feasibility of Selecting Patient-Specific Biologically Targeted Therapy With Sorafenib, Everolimus, Erlotinib or Dasatinib for Pediatric Patients With Refractory Or Recurrent Brain Tumors
Brief Title: Selecting Patient-Specific Biologically Targeted Therapy for Pediatric Patients With Refractory Or Recurrent Brain Tumors
Acronym: SEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, Sarah Leary, Associate Professor of Pediatrics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-9006
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Recurrent Childhood Brain Tumor
Keywords: Refractory; Recurrent; Brain; Tumor; Pediatric; Biologically Targeted Therapy; Sorafenib; Everolimus; Erlotinib; Dasatinib; Temozolomide; Etoposide
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — Immunohistochemistry; Temozolomide; Etoposide; etoposide phosphate; Sorafenib; Everolimus; Erlotinib Hydrochloride; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regimen B (Experimental): Depending on tumor biology testing, subjects assigned to Regimen B will receive:
  Temozolomide 150 mg/m2/dose daily PO on days 1-5, Etoposide 50 mg/m2/dose daily PO on days 1-12, and Everolimus 3 mg/m2/dose daily PO on days 1-28. Cycles will be repeated every 28 days for up to 12 cycles.
  Interventions: Device: Tumor biology testing; Drug: Temozolomide; Drug: Etoposide; Drug: Everolimus
- Regimen C (Experimental): Depending on tumor biology testing, subjects assigned to Regimen C will receive:
  Temozolomide 150 mg/m2/dose daily PO on days 1-5, Etoposide 50 mg/m2/dose daily PO on days 1-12, and Erlotinib 85 mg/m2/dose daily PO on days 1-28. Cycles will be repeated every 28 days for up to 12 cycles.
  Interventions: Device: Tumor biology testing; Drug: Temozolomide; Drug: Etoposide; Drug: Erlotinib
- Regimen D (Experimental): Depending on tumor biology testing, subjects assigned to Regimen D will receive:
  Temozolomide 150 mg/m2/dose daily PO on days 1-5, Etoposide 50 mg/m2/dose daily PO on days 1-12, and Dasatinib 60 mg/m2/dose BID PO on days 1-28. Cycles will be repeated every 28 days for up to 12 cycles.
  Interventions: Device: Tumor biology testing; Drug: Temozolomide; Drug: Etoposide; Drug: Dasatinib
- Regimen A (Experimental): Depending on tumor biology testing, subjects assigned to Regimen A will receive:
  Temozolomide 150 mg/m2/dose daily PO on days 1-5, Etoposide 50 mg/m2/dose daily PO on days 1-12, and Sorafenib 150 mg/m2/dose BID PO on days 1-28. Cycles will be repeated every 28 days for up to 12 cycles.
  Interventions: Device: Tumor biology testing; Drug: Temozolomide; Drug: Etoposide; Drug: Sorafenib

INTERVENTIONS:
Device: Tumor biology testing — Tumor biology studies will be performed in a CLIA-approved clinical pathology laboratory using standard procedures. Immunohistochemical (IHC) testing will be performed on formalin fixed tumor obtained at the time of diagnosis and/or relapse. Results will be interpreted by a qualified pediatric pathologist and will be scored on a scale of 0 to 4+ commenting on both percentage of positive cells and intensity of staining. Results will further be reported as a binary result (positive/negative). If more than one tumor specimen is available from different surgical procedures (e.g. initial diagnosis and relapse), the results from the relapse specimen will be prioritized. Results will determine kinase inhibitor treatment arm assignment which will be administered in addition to the "best available" combination of low-dose oral cytotoxic agents, including temozolomide and etoposide.
  Other Names: IHC Testing; Immunohistochemical Screening; Immunohistochemical Test; Tumor Markers
Drug: Temozolomide — Temozolomide combined with Etoposide is considered the "best available" combination of low-dose oral cytotoxic agents for patients with refractory or recurrent CNS tumors.
  Other Names: Temodar; Temodal; Temcad
Drug: Etoposide — Etoposide combined with Temozolomide is considered the "best available" combination of low-dose oral cytotoxic agents for patients with refractory or recurrent CNS tumors.
  Other Names: Etopophos; Vepesid
Drug: Sorafenib — Sorafenib is a broad-spectrum kinase inhibitor.
  Other Names: Nexavar
  Arms: Regimen A
Drug: Everolimus — Everolimus is an mTOR pathway inhibitor.
  Other Names: Zortress; Certican
  Arms: Regimen B
Drug: Erlotinib — Erlotinib is a tyrosine kinase inhibitor of the ERBB family of proteins.
  Other Names: Tarceva
  Arms: Regimen C
Drug: Dasatinib — Dasatinib is a broad spectrum SRC inhibitor.
  Other Names: Sprycel
  Arms: Regimen D

SUMMARY:
This research study is a Feasibility clinical trial. In this trial, researchers are trying to figure out whether a medication can be chosen based on rapid testing done on tumor tissue. Information from a feasibility or pilot trial will hopefully help researchers plan larger trials in the future to determine the effect of this therapy.

DETAILED DESCRIPTION:
This research study will assign a specific drug treatment based on lab tests performed on the participant's tumor from tumor tissue taken from a biopsy done when he/she was first diagnosed or if taken when he/she relapsed or progressed. All participants will get Temozolomide and Etoposide to start. Then depending on review of the participant's tumor tissue he/she will also receive one of the following: Sorafenib, Everolimus, Erlotinib, or Dasatinib.

The purpose of this research study is to learn about the feasibility of obtaining and using information from studies done on tumor tissue in order to help make treatment decisions for patients with relapsed or refractory pediatric brain tumors. The investigators also want to find out the effects this therapy has on the participant and the participant's brain tumor.

ELIGIBILITY:
Inclusion Criteria:

Patients must have histological confirmation of a brain tumor at diagnosis or relapse for all tumors.

There must be documented progression or recurrence of disease by MRI imaging or CSF studies since completion of last tumor-directed medical therapy. Patients may have had surgical resection or radiation of tumor, and need not have measurable or evaluable disease at study entry.

Patient's current disease state must be one for which there is no known curative therapy.

Age greater than 1 month and less than 30 years at the time of enrollment.

BSA greater than 0.3 m2 at the time of enrollment.

Karnofsky >/= 50% for patients > 16 years of age, and Lansky >/= 50% for patients </= 16 years of age.

* Neurologic deficits in patients with CNS tumors must have been relatively stable for a minimum of 7 days.
* Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Adequate bone marrow function including:

* ANC > 750
* Platelet count > 100,000/uL without platelet transfusion within the past 7 days

Adequate renal function defined as creatinine within normal range for age or calculated GFR > 100 ml/min/1.73 m2.

Adequate liver function defined as Bilirubin < 1.5 x upper limit of normal and ALT < 2.5 x upper limit of normal.

Adequate CNS function:

* Patients with known seizure disorder must have seizures adequately controlled with non-enzyme inducing antiepileptic medications
* No increase in steroid dose within the past 7 days.

Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy:

* Myelosuppressive chemotherapy: Must not have received within 3 weeks of entry onto this study (6 weeks if prior nitrosourea).
* Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor, 14 days for longacting (e.g. PEG-filgrastim)
* Biologic (anti-neoplastic agent): At least 7 days or 3 half-lives (whichever is longer) since the completion of therapy with a biologic agent.
* Radiation therapy: ≥ 12 weeks must have elapsed from craniospinal radiation; ≥ 2 weeks must have elapsed from focal radiation.
* Surgery: > 3 weeks from major surgery. If recent craniotomy, adequate wound healing must be determined by neurosurgical team prior to starting study therapy.
* Autologous Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and ≥ 4 weeks must have elapsed.

All patients and/or a legal guardian must sign institutionally approved written informed consent document.

Exclusion Criteria:

Patients who are breastfeeding, pregnant or refuse to use an effective form of birth control are excluded. Abstinence is considered an effective form of birth control.

Patients with uncontrolled infection are excluded.

Patients with known bleeding disorders or more than punctate intratumoral hemorrhage are excluded.

Patients receiving other anti-neoplastic agents are excluded.

Patients on enzyme-inducing anticonvulsive agents are excluded.

Patients requiring strong CYP3A4 inducers or inhibitors are excluded.

Patients requiring anticoagulation or with uncontrolled bleeding are excluded.

Patients on steroids for symptom management must be on a stable dose over the 7 days prior to study enrollment.

Patients within 1 year of allogeneic stem cell transplant, patients with active GVHD or requiring immunosuppression are excluded.

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 3 years
  It will be considered feasible to obtain individual biologic testing if at least 80% of patients receive results of biology studies within two weeks of study enrollment.
  It will be considered feasible to treat patients based on biologic testing if at least and 50% of patients who consent for biology testing start therapy with one of four regimens within four weeks of study enrollment.

SECONDARY OUTCOMES:
Efficacy | 3 years
  Efficacy endpoint for patients with evaluable or measurable disease will be best objective response (CR, PR, SD or PD) measured by MRI imaging.
Survival | 3 years
  Survival endpoints will be estimated including time to progression as well as progression-free and overall survival rates at the 6 month, 1 year and 2 year time point from start of study treatment.
Toxicity | 3 years
  Toxicity endpoints will be descriptive and include grading of patient toxicity according to the National Cancer Institute common terminology criteria for adverse events (CTCAE version 4.0). This study is not intended or powered to compare toxicity between treatment arms. The tolerability of selected therapy with the addition of a kinase inhibitor will be described for all patients as a group.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah ES Leary, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States